CLINICAL TRIAL: NCT00114478
Title: Randomized Controlled Trial of Epinephrine and Albuterol in Bronchiolitis
Brief Title: Trial of Epinephrine and Albuterol in Bronchiolitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMC03034
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; disposition; pediatric; epinephrine; albuterol
MeSH Terms: conditions — Bronchiolitis | interventions — Epinephrine; Albuterol

INTERVENTIONS:
Drug: Epinephrine
Drug: albuterol (salbutamol)

SUMMARY:
The purpose of this study is to see which of the two most common drugs used to treat bronchiolitis works better. A child's participation in this study is expected to last less than 4 hours. Approximately 600 patients will be recruited to participate in this study at Kern Medical Center (KMC).

Bronchiolitis is a very common lung infection in babies. There are many drugs used to treat this disease but nobody knows which one, if any, works the best. Two of the most commonly used drugs are albuterol and epinephrine. These are both drugs given during breathing treatments with oxygen and a mask. We are doing this study to see which of these drugs works better or if they are both equally good. The study works as follows: after the consent process the baby gets three treatments.

* Nebulizer 1 (Treatment)
* Treatment + 30 minutes (approximately) Nebulizer 2
* Treatment + 60 minutes (approximately) Nebulizer 3
* Treatment + 120 minutes (approximately)

The baby will be reevaluated and either discharged home or revert to standard therapy. If the baby is discharged directly from the emergency department (E.D.), we will call you in three days time to see how he/she is doing.

DETAILED DESCRIPTION:
Double blind RCT. Primary outcome measure is admission defined as actual admission or discharge with unscheduled return leading to admission within 72 hours. Secondary endpoints include change in severity of illness and response of respiratory parameters to treatment.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of bronchiolitis

Exclusion Criteria:

* Age greater than 18 months
* Disease too mild to warrant any treatment
* Emergent intubation on arrival at the ED
* Participation within another study within 30 days
* Refusal of informed parental consent

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600
Dates: Start 2003-11; Study Completion 2006-05

PRIMARY OUTCOMES:
Successful hospital discharge at three days

SECONDARY OUTCOMES:
Improvement in severity of disease score
Improvement in respiratory status

CONTACTS AND LOCATIONS:
Overall Officials: Paul Walsh, Paul Walsh, MD MSc(peds), Principal Investigator — Kern Medical Center, David Geffen School of Medicine, UCLA; Paul Walsh, Principal Investigator — Research Director, Emergency Medicine
Locations (1):
- Kern Medical Center, Bakersfield, California, United States

REFERENCES:
- [Background] Walsh P, Rothenberg SJ, O'Doherty S, Hoey H, Healy R. A validated clinical model to predict the need for admission and length of stay in children with acute bronchiolitis. Eur J Emerg Med. 2004 Oct;11(5):265-72. doi: 10.1097/00063110-200410000-00005. PMID 15359199
- [Derived] Walsh P, Caldwell J, McQuillan KK, Friese S, Robbins D, Rothenberg SJ. Comparison of nebulized epinephrine to albuterol in bronchiolitis. Acad Emerg Med. 2008 Apr;15(4):305-13. doi: 10.1111/j.1553-2712.2008.00064.x. PMID 18370982
- See also: Research assistant site for this study. Restricted access. — http://groups.yahoo.com/group/kmcemrap